CLINICAL TRIAL: NCT03526081
Title: Absorption, Metabolism and Excretion of Apigenin and Apigenin Glycosides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 429275-10
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: flavone; ADME; apigenin; parsley; chamomile; polyphenols
MeSH Terms: interventions — Chamomile extract; Apigenin

STUDY DESIGN:
Intervention Model Description: Cross-over dietary intervention study in healthy young adult males
Who Masked: Investigator
Masking Description: Investigator doing data analysis and statistical analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chamomile Tea (Experimental): Chamomile Tea in 300mL hot water
  Interventions: Other: Chamomile Tea
- Parsley based drink (Experimental): 3.2 g dried parsley in 300mL hot water
  Interventions: Other: Parsley based drink
- Parsley Yogurt (Experimental): 3.2 g dried parsley in 100g plain yogurt
  Interventions: Other: Parsley Yogurt
- Apigenin (Experimental): Apigenin capsule mixed with 300mL hot water
  Interventions: Other: Apigenin
- Parsley-based drink (II) (Experimental): 3.2 g of dried parsley in 300 ml of hot water
  Interventions: Other: Parsley-based drink (II)

INTERVENTIONS:
Other: Chamomile Tea — Chamomile Tea in 300mL hot water
  Arms: Chamomile Tea
Other: Parsley based drink — 3.2 g dried parsley in 300mL hot water
  Arms: Parsley based drink
Other: Parsley Yogurt — 3.2 g dried parsley in 100g plain yogurt
  Arms: Parsley Yogurt
Other: Apigenin — Apigenin capsule mixed with 300mL hot water
  Arms: Apigenin
Other: Parsley-based drink (II) — 3.2 g dried parsley in 300mL hot water
  Arms: Parsley-based drink (II)

SUMMARY:
Probe dietary intervention study in healthy young adult males to evaluate the concentration of apigenin derived metabolites in plasma and urine after single acute intakes of different apigenin-containing test materials.

DETAILED DESCRIPTION:
Flavonoids, including the sub groups of Flavones (FO) are plant-derived compounds commonly present in the human diet. Examples of FO-containing foods and beverages are parsley, celery, and chamomile. The study described below will provide initial information of apigenin derived metabolites in humans. The investigators suggest the information that will be obtained from the outlined work will be particularly timely given increasing interest in the putative health effects of FO intake in humans.

This study consisted of two parts. The first part consisted of a probe study in which the investigators investigated the absorption and metabolism from four flavone-containing test products. The second phase investigated absorption and metabolism after the intake of a flavone-containing parsley drink.

ELIGIBILITY:
Inclusion Criteria:

* No prescription medications
* BMI 18.5 - 29.9 kg/m2
* Weight ≥ 110 pounds
* previously consumed cocoa, peanut, parsley, celery and chamomile products with no adverse reactions

Exclusion Criteria:

* Adults unable to consent
* Prisoners
* Non-English speaking
* BMI ≥ 30 kg/m2
* Performing vigorous physical activity (i.e. more than 6 metabolic equivalence of task (MET) as defined by Centers for Disease Control and Prevention (CDC) and American College of Sports Medicine (ACSM) guidelines) for more than 3 days a week
* Dietary allergies including those to nuts, cocoa and chocolate products, parsley, celery and chamomile.
* Active avoidance of coffee and caffeinated soft drinks
* Under current medical supervision
* A history of cardiovascular disease, stroke, renal, hepatic, or thyroid disease
* History of clinically significant depression, anxiety or other psychiatric condition
* History of Raynaud's disease
* History of difficult blood draws
* Indications of substance or alcohol abuse within the last 3 years
* Current use of herbal, plant or botanical supplements (multi-vitamin/mineral supplements are allowed)
* Blood Pressure > 140/90 mm Hg
* GI tract disorders, previous GI surgery (except appendectomy)
* Self-reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food, potentially leading to bloating, cramping or gas)
* Diarrhea within the last 3 months, or antibiotic intake within the last 3 months
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, on a weight loss diet or individuals following diets with significant deviations from the average diet
* Metabolic panel and cholesterol results or complete blood counts that are outside of the normal reference range and are considered clinically relevant by the study physician
* Cold, flu, or upper respiratory condition at screening
* Currently participating in a clinical or dietary intervention study

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Flavone metabolites in plasma | before to 6 h post test material intake
  Concentration of flavone metabolites in plasma
Flavone metabolites in urine | 12 h before to 24 h post test material intake
  Amount of flavone metabolites excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — UC Davis; Javier I Ottaviani, PhD, Study Director — Mars, Inc.
Locations (2):
- United States (2):
  - Ragle Human Nutrition Research Center, Department of Nutrition at UC Davis, Davis, California
  - UC Davis, Davis, California

IPD SHARING:
Plan to Share IPD: Yes
Only researchers listed in the protocol and approved by the IRB will have access to IPD.

REFERENCES:
- [Background] Schroeter H, Heiss C, Spencer JP, Keen CL, Lupton JR, Schmitz HH. Recommending flavanols and procyanidins for cardiovascular health: current knowledge and future needs. Mol Aspects Med. 2010 Dec;31(6):546-57. doi: 10.1016/j.mam.2010.09.008. Epub 2010 Sep 18. PMID 20854838
- [Background] Ottaviani JI, Momma TY, Kuhnle GK, Keen CL, Schroeter H. Structurally related (-)-epicatechin metabolites in humans: assessment using de novo chemically synthesized authentic standards. Free Radic Biol Med. 2012 Apr 15;52(8):1403-12. doi: 10.1016/j.freeradbiomed.2011.12.010. Epub 2011 Dec 23. PMID 22240152
- [Background] Koster H, Halsema I, Scholtens E, Knippers M, Mulder GJ. Dose-dependent shifts in the sulfation and glucuronidation of phenolic compounds in the rat in vivo and in isolated hepatocytes. The role of saturation of phenolsulfotransferase. Biochem Pharmacol. 1981 Sep 15;30(18):2569-75. doi: 10.1016/0006-2952(81)90584-0. No abstract available. PMID 6946775
- [Background] McCullough ML, Chevaux K, Jackson L, Preston M, Martinez G, Schmitz HH, Coletti C, Campos H, Hollenberg NK. Hypertension, the Kuna, and the epidemiology of flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S103-9; discussion 119-21. doi: 10.1097/00005344-200606001-00003. PMID 16794446
- [Background] Heiss C, Kleinbongard P, Dejam A, Perre S, Schroeter H, Sies H, Kelm M. Acute consumption of flavanol-rich cocoa and the reversal of endothelial dysfunction in smokers. J Am Coll Cardiol. 2005 Oct 4;46(7):1276-83. doi: 10.1016/j.jacc.2005.06.055. PMID 16198843
- [Derived] Borges G, Fong RY, Ensunsa JL, Kimball J, Medici V, Ottaviani JI, Crozier A. Absorption, distribution, metabolism and excretion of apigenin and its glycosides in healthy male adults. Free Radic Biol Med. 2022 May 20;185:90-96. doi: 10.1016/j.freeradbiomed.2022.04.007. Epub 2022 Apr 20. PMID 35452808